CLINICAL TRIAL: NCT04142229
Title: A Randomized Crossover Comparison of Artificial Pancreas vs. Sensor Augmented Pump/Predictive Low Glucose Suspend With Different Stress Assessments in the Outpatient Setting for Patients With Type 1 Diabetes
Brief Title: Artificial Pancreas With Different Stress Assessments in the Outpatient Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Mayo Clinic (Other); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19-006965
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; automated insulin delivery; artificial pancreas; stress
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Automated Insulin Delivery (Experimental): Participants will use the Automated Insulin Delivery (AID) iAPS system for 2 weeks in the outpatient setting, and come to the clinical center twice for supervised stress assessments.
  Interventions: Device: iAPS
- SAP/PLGS (Active Comparator): Participants will use their home pump with a CGM sensor (sensor augmented pump) or in Predictive Low Glucose Suspend (PLGS) mode if their home pump supports this mode, for 2 weeks in the outpatient setting, and come to the clinical center twice for supervised stress assessments.
  Interventions: Other: Sensor-Augmented Pump

INTERVENTIONS:
Device: iAPS — The AID system (iAPS) is comprised of an insulin pump, a Dexcom G6 continuous glucose monitoring sensor, and a smart phone that contains the algorithm and communicates with the other devices.
  Arms: Automated Insulin Delivery
Other: Sensor-Augmented Pump — Subjects will use their home insulin pump and a Dexcom G6 continuous glucose monitoring sensor.
  Arms: SAP/PLGS

SUMMARY:
This feasibility study is a randomized crossover trial that will compare the efficacy and safety of an automated insulin delivery (AID) system in patients with type 1 diabetes using a Model Predictive Control (MPC) algorithm versus sensor augmented pump therapy (SAP)/Predictive Low Glucose Suspend (PLGS), and will include different stress induction and assessments over a 4 week period.

DETAILED DESCRIPTION:
Eligible participants will be randomly assigned to one of two treatment arms: 1) AID for two weeks and SAP/PLGS for two weeks , or 2) SAP/PLGS for two weeks and AID for two weeks. During the 4-week trial, subjects will wear the Empatica E4 wristband every day to record electrodermal activity, accelerometer and heartrate data. Subjects will also complete logbooks to record activity and stress. During each two-week period, subjects will come to the clinical center twice for stress induction tests in a medically supervised setting.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year and using insulin for at least 1 year
* Using an insulin pump for at least 3 months at the time of screening. Insulin pump use includes use of automated features, to include predictive or threshold low-glucose suspend or hybrid closed-loop with or without a Dexcom sensor.
* Familiarity and use of a carbohydrate ratio for meal boluses.
* Age ≥18.0 years old
* HbA1c < 10.5%, as performed by point of care or central laboratory testing. HbA1c will be assessed at the screening visit, or if already completed within 2 weeks of the screening visit, the prior lab value may be used in lieu of repeating this assessment.
* For females, not currently known to be pregnant. If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study and up to one month afterwards. A negative serum or urine pregnancy test will be required for all females of child-bearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
* Willingness to switch home pump to PLGS or full manual mode if using hybrid - Investigator has confidence that the participant can successfully operate all study devices and is capable of adhering to the protocol.
* Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use no other insulin besides lispro (Humalog) or aspart (Novolog) during the study.
* Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial.

Exclusion Criteria:

* Use of an unapproved closed-loop insulin delivery system within 2 weeks before screening or during the study is not allowed.
* Have a blood pressure at screening outside the range of 160 mmHg systolic blood pressure and/or greater than 100 mmHg for diastolic blood pressure (if repeated measurements are within this range, the patient may be included in the study)
* Have coronary artery disease that is not stable with medical management, including unstable angina, angina that prevents moderate exercise despite medical management, or within the last 12 months before screening a history of myocardial infarction, percutaneous coronary intervention, enzymatic lysis of a presumed coronary occlusion, or coronary artery bypass grafting
* Concurrent use of Afrezza or any non-insulin glucose-lowering agent other than metformin (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas).
* Hemophilia or any other bleeding disorder
* A condition, which in the opinion of the investigator or designee, would put the participant or study at risk, to include:

  * Pregnancy, or planning pregnancy within 1 month of completing the clinical trial.
  * Allergy or hypersensitivity to hydrocortisone, or any component of the formulation
  * Presence of a known adrenal disorder
  * Systemic fungal infections
  * Active infection of any kind, or at risk of infection (susceptibility to infection) from known immunosuppression or underlying immunosuppressed condition
  * Idiopathic thrombocytopenia purpura (ITP)
  * Varicella
  * Glaucoma or other chronic ocular condition that could be adversely affected by steroids (e.g., cataracts, increased ocular pressure from other causes, exophthalmos)
  * Hypertension requiring treatment with one or more antihypertensive medications
  * Congestive heart failure
  * Current treatment for a seizure disorder
  * Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation, including subjects not able to read or write
  * Known coronary artery disease
  * Active gastroparesis
  * Cystic fibrosis
  * Uncontrolled thyroid disease (TSH undetectable or > 10 mIU/L)
  * Known abuse of alcohol
  * A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol
  * Current use of a beta blocker medication
  * Laboratory results:

    * HbA1c > 10.5%
    * Abnormal liver or renal function (Transaminase >2 times the upper limit of normal, creatinine> 1.5 mg/dL)
    * Labs drawn at screening visit or within three months prior to screening (for other purposes) will suffice for enrollment purposes
  * Subject has skin conditions that, in the determination of the investigator, would preclude wearing the study devices (infusion set and sensor), in the abdomen. Examples include but are not limited to: psoriasis, burns, scaring, eczema, tattoos, and significant hypertrophy at sites of device wear; any known allergy to medical adhesives.
  * Currently on long-term treatment using prednisone or other steroid
  * If subject had been on short term treatment of prednisone, defer enrollment until underlying condition and prednisone treatment have resolved.
  * Allergy to study drug, food or other study material.
  * Clinically significant physical examination, laboratory test, or vital sign abnormality.
  * Exposure to any investigational drug within 30 days.
  * History of malignancy within the 5 years before screening (other than basal cell carcinoma).
* Participation in another pharmaceutical or device trial at the time of enrollment or during the study
* Having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Time in target glucose range | 4 weeks
  Time in target glucose range 70-180 mg/dL measured by CGM to determine safety and efficacy of the integrated system

SECONDARY OUTCOMES:
Change in glucose levels with stress induction | 4 weeks
  Change in glucose levels with stress induction sessions (mg/dL)
Change in insulin requirements with stress induction | 4 weeks
  Change in insulin requirements with stress induction sessions (units of insulin)
EDA stress detection | 4 weeks
  Analysis of EDA to verify stress detection and correlation to glucose changes, both during the stress sessions and in the outpatient setting
Postprandial Time in Target Range | 4 weeks
  Percent time within the target range of 70-180 mg/dl postprandial within 5 hours following meals
Glucose < 70 mg/dL | 4 weeks
  Percent time GGM glucose < 70 mg/dL
Glucose < 54 mg/dL | 4 weeks
  Percent time GGM glucose < 54 mg/dL
Glucose > 180 mg/dL | 4 weeks
  Percent time GGM glucose > 180 mg/dL
Glucose > 250 mg/dL | 4 weeks
  Percent time GGM glucose > 250 mg/dL
Serious adverse events (SAE) | 4 weeks
  The total number of serious adverse events during the clinical trial
Serious adverse device events (SADE) | 4 weeks
  The total number of serious adverse events related to the study device use during the clinical trial
Adverse device effects (ADE) | 4 weeks
  The total number of adverse device effects (ADE) during the clinical trial
Unanticipated adverse device effects (UADE) | 4 weeks
  The total number of unanticipated adverse device effects (UADE) during the clinical trial
Salivary cortisol assessment | 4 weeks
  Salivary cortisol assessment (nmol/l) during psychologic and physiologic stress induction
Empatica device-based assessment of psychologic and physiologic stress | 4 weeks
  EDA Measurement of psychologic and physiologic stress from the Empatica E4 Watch
Trier Social Stress Test (TSST) | 4 weeks
  Trier Social Stress Test (TSST) score at end of each test induction
Socially evaluated cold-pressor test (SECPT) | 4 weeks
  Socially evaluated cold-pressor test (SECPT) score at end of each test induction

OTHER OUTCOMES:
Closed-Loop Active Time | 2 weeks
  Percent time (hours/day) of closed-loop use during the two weeks of iAPS use
Sensor Use Time | 4 weeks
  Total hours of CGM sensor use time during both use of SAP/PLGS and when using the iAPS
Device Issues | 4 weeks
  Total number of devices issues during the clinical trial
Total daily insulin use | 4 weeks
  Total daily insulin use (units/day) during both use of SAP/PLGS and when using the iAPS
Total basal insulin use | 4 weeks
  Total daily basal insulin use (units/day) during both use of SAP/PLGS and when using the iAPS
Total bolus insulin use | 4 weeks
  Total daily bolus insulin use (units/day) during both use of SAP/PLGS and when using the iAPS
Questionnaire Score | 2 weeks
  Questionnaire before and after AID use to assess technology acceptance, fear of hypoglycemia, diabetes associated distress (Likert Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Yogish Kudva, MBBS, Principal Investigator — Mayo Clinic; Eyal Dassau, PhD, Principal Investigator — Harvard University; Jordan Pinsker, MD, Principal Investigator — Sansum Diabetes Research Institute
Locations (2):
- United States (2):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pinsker JE, Deshpande S, McCrady-Spitzer S, Church MM, Kaur RJ, Perez J, Desjardins D, Piper M, Reid C, Doyle FJ 3rd, Kudva YC, Dassau E. Use of the Interoperable Artificial Pancreas System for Type 1 Diabetes Management During Psychological Stress. J Diabetes Sci Technol. 2021 Jan;15(1):184-185. doi: 10.1177/1932296820948566. Epub 2020 Aug 12. No abstract available. PMID 32783473
- [Derived] Kaur RJ, Deshpande S, Pinsker JE, Gilliam WP, McCrady-Spitzer S, Zaniletti I, Desjardins D, Church MM, Doyle Iii FJ, Kremers WK, Dassau E, Kudva YC. Outpatient Randomized Crossover Automated Insulin Delivery Versus Conventional Therapy with Induced Stress Challenges. Diabetes Technol Ther. 2022 May;24(5):338-349. doi: 10.1089/dia.2021.0436. Epub 2022 Apr 25. PMID 35049354